CLINICAL TRIAL: NCT02172001
Title: A Phase III, Randomised, Double-blind, Comparative Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Against Placebo in Subjects With Iron Deficiency Anaemia and Who Are Intol-erant or Unresponsive to Oral Iron Therapy
Brief Title: A Randomized, Double-blind, Comparative Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Against Placebo
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study design not adequate
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-Monofer-IDA-02
Record Dates: First submitted 2014-06-21; First posted 2014-06-24 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-03

CONDITIONS: Iron Deficiency Anemia
Keywords: IDA; Iron deficiency; iron deficiency anemia and who are intolerant or unresponsive to oral iron therapy
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — iron isomaltoside 1000

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron isomaltoside 1000 (Experimental): Iron isomaltoside 1000. Dose: 1000 mg, 1500 mg or 2000 mg
  Interventions: Drug: Iron isomaltoside 1000
- Placebo (NaCl 0,9%) (Placebo Comparator): Sodium Chloride. Dose: 100 ml or 5 ml
  Interventions: Drug: Natrium Chloride 0,9%

INTERVENTIONS:
Drug: Iron isomaltoside 1000
  Arms: Iron isomaltoside 1000
Drug: Natrium Chloride 0,9% — 100 ml or 5 ml
  Arms: Placebo (NaCl 0,9%)

SUMMARY:
The primary objective of the study is to evaluate and compare the effect of iron isomaltoside 1000 to placebo in its ability to increase haemoglobin (Hb) in subjects with IDA when oral iron preparations are ineffective or cannot be used.

DETAILED DESCRIPTION:
IDA is highly prevalent in subjects and can have a substantial medical and quality of life (QoL) burden on the subjects and the treatment of these subjects includes replenishing lost iron. Oral iron administration is often used in the clinical practice at many clinics; however, oral iron may not be tolerated by all subjects. Hence, there is a need for an alternative iron treatment in subjects, who do not tolerate oral iron.

This study is planned to compare the efficacy and safety of iron isomaltoside 1000 with placebo in subjects with IDA and who are intolerant or unresponsive to oral iron therapy..

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years having IDA caused by different aetiologies* such as ab-normal uterine bleeding, gastrointestinal diseases (e.g. inflammatory bowel disease), cancer, preoperative anaemia (e.g. orthopaedic surgery), and other conditions leading to IDA and with a documented history of intolerance or unresponsiveness to oral iron therapy** for at least one month*** prior to study enrolment
2. Hb < 11 g/dL
3. TSAT < 20 %
4. S-ferritin < 100 ng/mL
5. Willingness to participate and signing the informed consent form (ICF)

Exclusion Criteria:

1. Hb < 6 g/dL
2. Anaemia predominantly caused by factors other than IDA (e.g. anaemia with untreat-ed vitamin B12 or folate deficiency, haemolytic anaemia)
3. Iron overload or disturbances in utilisation of iron (e.g. haemochromatosis and hae-mosiderosis)
4. Decompensated liver cirrhosis or active hepatitis (ALAT > 3 times upper limit of normal)
5. Active acute or chronic infections (assessed by clinical judgement supplied with white blood cells (WBC) and C-reactive protein (CRP))
6. Body weight < 50 kg
7. Pregnant or nursing women. In order to avoid pregnancy, women of childbearing po-tential have to use adequate contraception (e.g. intrauterine devices, hormonal contra-ceptives, or double barrier method) during the whole study period and 7 days after the last dosing
8. History of multiple allergies
9. Known hypersensitivity to parenteral iron or any excipients in the investigational drug products
10. Erythropoietin treatment within 8 weeks prior to the screening visit
11. Other intravenous (IV) iron treatment or blood transfusion within 4 weeks prior to the screening visit
12. Participation in any other interventional clinical study within 3 months prior to the screening
13. Any other medical condition that, in the opinion of Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study, e.g. uncontrolled hypertension, unstable ischemic heart disease, or uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an Hb increase of ≥ 2 g/dL from baseline at any time from week 1 to week 5 | Week 1 to 5

SECONDARY OUTCOMES:
Time to Hb ≥ 2 g/dL | Week 1 to 5

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore, Maryland, United States